CLINICAL TRIAL: NCT03642977
Title: DNA and RNA Viruses of the Blood Virome of Allogeneic Hematopoietic Stem Cell Transplant Recipients: a Longitudinal Observational Study During a One-year Period After Transplantation - the Geneva Blood Virome Project (GeBVir)
Brief Title: DNA and RNA Viruses of the Blood Virome of Allogeneic Hematopoietic Stem Cell Transplant Recipients
Acronym: GeBVir
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Prof Laurent Kaiser (Unknown); Dr Samuel Cordey (Unknown); Dr Stavroula Masouridi-Levrat (Unknown); Prof Christian Van Delden (Unknown); Prof Yves Chalandon (Unknown); Dr Dionysios Neofytos (Unknown); Dr Federico Simonetta (Unknown); Dr Diem-Lan Vu Cantero (Unknown)
Responsible Party: Principal Investigator, Marie-Céline Zanella, Principal investigator, University Hospital, Geneva
Other Study IDs: Protocol 2017-01304
Record Dates: First submitted 2018-07-30; First posted 2018-08-22 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Hematopietic Stem Cell Transplantation; Blood Virome; RNA Virus Infections; DNA Virus Infections
Keywords: Longitudinal study; Real time PCR
MeSH Terms: conditions — RNA Virus Infections; DNA Virus Infections | interventions — DNA, B-Form

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic HSCT recipients: Adult patients receiving allogeneic hematopoietic stem cell transplant (HSCT) at University Hospitals of Geneva and who are enrolled in the "Cohort of infectious disease in hematopoietic stem cell transplant patients".
  Interventions: Diagnostic Test: Real time PCR and RT-PCR for DNA and RNA viral species

INTERVENTIONS:
Diagnostic Test: Real time PCR and RT-PCR for DNA and RNA viral species — Qualitative and quantitative real time PCR and RT-PCR assays will be performed on hematopoietic stem cell transplant recipients' plasma samples collected at five specific time points over a one-year period after transplantation (the day of transplantation (D0), 30 days (D30), 3 months (M3), 6 months (M6) and one year (Y1) after transplantation), for the screening of a selection of at least 21 DNA and RNA viruses (belonging to the Herpesviridae, Polyomaviridae, Adenoviridae, Parvoviridae, Anelloviridae, Picornaviridae and Flaviviridae families).

SUMMARY:
The Geneva Blood Virome Project is a longitudinal observational study. The main objective is to describe the kinetics of the plasmatic viral load of a selection of at least 21 DNA and RNA viruses of the blood virome in allogeneic hematopoietic stem cell transplant recipients, over a one-year period after transplantation. Secondary objectives are: 1) to assess the prevalence of DNA and RNA viruses plasmatic detections and co-detections, 2) to assess the cumulative incidence of DNA and RNA viruses plasmatic detection. The population of the study consists in adult patients receiving allogeneic stem cell transplantation at the University Hospitals of Geneva, enrolled in an already existing monocentric cohort, and for which clinical specimens are collected and stored at the time and after transplantation. The investigators plan to include 120 patients whose plasma samples are collected from March 2017 and to systematically use plasma samples collected on the day of transplantation and several time points after transplantation to screen DNA and RNA viruses by qualitative and quantitative real-time PCR and RT-PCR.

DETAILED DESCRIPTION:
The Geneva Blood Virome Project is a longitudinal observational study. The main objective is to describe the kinetics of the plasmatic viral load of a selection of at least 21 DNA and RNA viruses of the blood virome (Herpesviridae Polyomaviridae, Adenoviridae, Parvoviridae, Anelloviridae, Picornaviridae and Flaviviridae) in allogeneic hematopoietic stem cell transplant recipients, over a period of one year after transplantation. These DNA and RNA viruses can be responsible of acute infections, chronic infections or reactivations after transplantation. Secondary objectives are : 1) to assess the prevalence of DNA and RNA viruses plasmatic detections and co-detections at pre-specified time-points, 2) to assess the cumulative incidence of DNA and RNA viruses plasmatic detection at pre-specified time-points. The population of the study consists in adult patients receiving allogeneic stem cell transplantation at the University Hospitals of Geneva and who are enrolled in an already existing monocentric cohort named "Cohort of infectious disease in hematopoietic stem cell transplant patients" and for which clinical specimens are collected and stored at the time and after transplantation. The investigators plan to include 120 patients whose plasma samples are collected from March 2017 and to systematically use plasma samples collected at 5 pre-specified time points (the day of transplantation, 30 days, 3 months, 6 months, and one year after transplantation) to perform qualitative and quantitative real-time r(RT)-PCR assays for the screening of DNA and RNA viruses. The definitive analysis of results should be done by the end of 2020.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving allogeneic stem cell transplantation since March 2017 at University Hospitals of Geneva
* Enrollment in the "Cohort of infectious disease in hematopoietic stem cell transplant patients"
* Signature of an informed consent form before transplantation

Exclusion Criteria:

* Absence of a signed informed consent form for the "Cohort of infectious disease in hematopoietic stem cell transplant patients".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving allogeneic stem cell transplantation at University Hospitals of Geneva and who are enrolled in an already existing monocentric cohort named "Cohort of infectious disease in hematopoietic stem cell transplant patients"
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Plasmatic viral load kinetics of DNA and RNA viruses | one-year period after transplantation
  Measurement of the plasmatic viral load of DNA and RNA viruses belonging to the Herpesviridae, Polyomaviridae, Adenoviridae, Parvoviridae, Anelloviridae, Picornaviridae and Flaviviridae families, with real time (RT-)PCR on plasma samples collected at pre-specified timepoints (the day of transplantation (D0), 30 days (D30), 3 months (M3), 6 months (M6) and one year (Y1) after transplantation) (expressed as fold-increase).

SECONDARY OUTCOMES:
Prevalence of plasmatic detection of DNA and RNA viruses | one-year period after transplantation
  Detection of DNA and RNA viruses using real time (RT-)PCR performed on plasma samples collected at pre-specified timepoints
Cumulative incidence of DNA and RNA viruses plasmatic detection | one-year period after transplantation
  Detection of DNA and RNA viruses using real time (RT-)PCR performed on plasma samples collected at pre-specified timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Céline Zanella, Principal Investigator — University Hospitals of Geneva; Laurent Kaiser, Principal Investigator — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided